CLINICAL TRIAL: NCT06951334
Title: Clinical Trial of Vildagliptin in Early Parkinson's Disease
Acronym: VERY-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhang Nu, Prof, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2024]746; FirstSunYetSen (Other: SunYetSen)
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
MeSH Terms: interventions — Vildagliptin; BID protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional medication plus Vildagliptin treatment group (Experimental): Traditional dopamine preparations combined with vildagliptin treatment
  Interventions: Drug: Vildagliptin 50 mg bid
- conventional medication treatment group (No Intervention): Only traditional dopamine preparations are used for treatment without additional intervention

INTERVENTIONS:
Drug: Vildagliptin 50 mg bid — Vildagliptin 50 mg bid for 12months
  Arms: Conventional medication plus Vildagliptin treatment group

SUMMARY:
Investigating the efficacy of Vildagliptin in delaying the progression of Parkinson's disease.

DETAILED DESCRIPTION:
Exploring the effectiveness and safety of vildagliptin in delaying the progression of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients aged 40 to 75 years who were diagnosed with Parkinson's disease according to the UK Brain Bank criteria within the past three years.

  2: Participants must have received an optimized and stable dopaminergic medication regimen (dopamine agonists, levodopa, or monoamine oxidase B [MAOB] inhibitors, or combinations of these medications) determined by the study site investigators for at least one month prior to the baseline initiation of the trial drug, with the expectation that the participants will be able to continue this regimen for at least six months.

  3: Sign the informed consent form

Exclusion Criteria:

* 1: The key exclusion criterion is a score of at least 3 on the Hoehn and Yahr scale (ranging from 1 to 5, with higher scores indicating more severe disability), which indicates that Parkinson's disease has led to at least mild to moderate bilateral motor involvement due to some postural instability.

  2: Presence of motor fluctuations or motor complications (or both).

  3: The presence of severe psychiatric disorders, such as severe (treatment-resistant) anxiety, depression, or schizophrenia, that cannot be effectively controlled by medication.

  4: Atypical or secondary Parkinsonism

  5: A score of 18 or lower on the Montreal Cognitive Assessment (MoCA) (range: 0 to 30, with a score of 26 or higher indicating normal cognitive function), indicating at least mild cognitive impairment.

  6: Diabetes mellitus (Type 1 and Type 2), as well as prior treatment with dipeptidyl peptidase-4 (DPP-4) inhibitors or glucagon-like peptide-1 (GLP-1) receptor agonists.

  7: Individuals with severe renal impairment (creatinine clearance <30 ml/min), active liver disease, history of drug or alcohol abuse, idiopathic pancreatitis, chronic pancreatitis, or a history of pancreatectomy.

  8: Individuals with a body mass index (weight in kilograms divided by the square of height in meters) less than 18.5, or those with a weight change exceeding 5 kilograms within the 3 months prior to screening.

  9: Currently participating in other relevant clinical trials involving pharmacological or surgical treatments.

  10: Other situations where the investigator believes that the subject is unable to participate in or cooperate with the entire assessment process of the clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in the third part of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) after 12 months of oral Vildagliptin treatment compared to baseline | baseline, pre-intervention；12 months，month 12
  MDS-UPDRS Part III mainly includes motor symptoms (total score 0-132 points), with scores ranging from 0 to 132 The higher the symptom, the more severe it is.